CLINICAL TRIAL: NCT04128852
Title: A Prospective, Single Arm, Single-center Study to Assess the Safety and Performance of MagnetOs Putty in Patients Undergoing Single/Two-level Lateral Lumbar Interbody Fusion
Brief Title: Post Marketing Clinical Follow up Study for MagnetOs Putty in Patients With Degenerative Disc Disease
Acronym: PROGRESS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: redirected funding
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Factory CRO (Industry); The London Clinic (Other); Kuros BioSciences B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAG-919-013
Record Dates: First submitted 2019-10-04; First posted 2019-10-16 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Disc Disease
Keywords: Spinal Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Single arm, single-center, post market surveillance study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MagnetOs Putty (Other): MagnetOs Putty will be applied according to the latest Instructions For Use (IFU) approved in Europe. Specifically, MagnetOs Putty will be used as bone void filler.
  Interventions: Device: MagnetOs Putty

INTERVENTIONS:
Device: MagnetOs Putty — MagnetOs Putty has a CE-mark (2115660CE01) as well as FDA 510(k) clearance (K171563/K181958).

SUMMARY:
This study is a post-marketing clinical follow-up study for MagnetOs Putty. MagnetOs Putty is a synthetic bone-like material which is routinely used by surgeons as a treatment for patients with degenerative disc disease who will undergo surgery for spinal fusion (extreme lateral interbody fusion (XLIF). MagnetOs Putty will be used according to the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by the patient.
2. Male or female patient ≥ 25 up to and including 75 years old.
3. Patients with degenerative disc disease with up to grade 1 spondylolisthesis and with leg pain requiring 1 to 3 level laminectomy and a single/two-level fusion (L2 - S1). Degenerative disc disease is defined by the presence of one or more of the following:

   1. instability (angulation ≥ 5 degrees or translation ≥ 3 mm on flexion/extension radiographs),
   2. osteophyte formation of facet joints or vertebral endplates,
   3. decreased disc height by > 2 mm, but dependent upon the spinal level,
   4. scarring/thickening of ligamentum flavum, annulus fibrosis or facet joint capsule,
   5. disc degeneration and/or herniation,
   6. facet degeneration,
   7. vacuum phenomenon.
4. Patients with an Oswestry Disability Index (ODI) score ≥ 30.
5. Patients with a Visual Analogue Scale (VAS) leg score ≥ 40.
6. Failed conservative treatment (physical therapy, bed rest, medications, spinal injections or transcutaneous electrical nerve stimulation) for a period of 6 months prior to study enrollment.

Exclusion Criteria:

Per the current Instruction For Use, MagnetOs Putty must not be used in the following clinical situations:

1. To treat conditions in which general bone grafting is not advisable.
2. In conditions where the surgical site may be subjected to excessive impact or stresses, including those beyond the load strength of fixation hardware (e.g. defect site stabilisation is not possible).
3. In case of significant vascular impairment proximal to the graft site.
4. In case of severe metabolic or systemic bone disorders that affect bone or wound healing.
5. In case of acute and chronic infections in the operated area (soft tissue infections; inflammation, bacterial bone diseases; osteomyelitis).
6. When intraoperative soft tissue coverage is not planned or possible.
7. In direct contact with the articular space.
8. In case of treatment with medication interfering with the calcium metabolism.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic interbody fusion by CT scan | 12 months
  The rate of interbody fusion assessed by CT-scan at Month 12. Radiographic fusion using CT-scan will be defined by an independent radiology expert at Month 12 post-surgery and determined by evidence of bridging trabeculae or continuous bony connection between superior and inferior vertebral body.

IPD SHARING:
Plan to Share IPD: No